CLINICAL TRIAL: NCT06175299
Title: Evaluating the Social Functions to Promote the Adherence and Reduce Social Isolation in Home-based Cognitive Training
Brief Title: Social Functions to Promote Home-based Cognitive Training
Acronym: DeepCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Zhe He, Principal Investigator, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FSU00004067
Record Dates: First submitted 2023-12-06; First posted 2023-12-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Adherence, Treatment; Social Isolation
Keywords: Cognition; Adherence; Social isolation
MeSH Terms: conditions — Treatment Adherence and Compliance; Social Isolation | interventions — 4-azido-7-phenylpyrazolo-(1,5a)-1,3,5-triazine; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Training with Social Function (Experimental): To promote adherence and reduce social isolation, participants will be asked to use home-based cognitive training program on a tablet for 30 minutes per day for 5 days a week for 1 month, then use it freely for another month. The cognitive training program has a chat function and a leadership board to allow interaction between participants.
  Interventions: Behavioral: Adherence Promotion With Person-centered Technology (APPT) System with Social Functions

INTERVENTIONS:
Behavioral: Adherence Promotion With Person-centered Technology (APPT) System with Social Functions — The system has seven games for cognitive training and two social interactions functions: a chat function and a leaderboard function.

SUMMARY:
This study will examine whether among older adults social interaction functions in a home-based cognitive training program can better support adherence to training and reduce social isolation.

DETAILED DESCRIPTION:
The goal of this project is to conduct a pilot study to test the feasibility of two new features, a chat function and a leaderboard function, to encourage social interactions and support adherence to cognitive training protocols (mental exercises delivered via a tablet) over a period of time (2 months), and uncover individual difference factors that can predict poor adherence in the future and social interactions in the game. Even effective cognitive interventions may fail if individuals do not adhere to them for an extended period. This project will compare cognitive training games with chat function and leaderboard in reducing social isolation and improving adherence to the training, compared to an external control group using a generic reminder system delivered via smartphone text messages to promote adherence. The ultimate goal, as effective technology-based interventions to improve cognition become available, is to help support their benefit for older adults by maximizing long-term adherence.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Normal or corrected to normal visual acuity
* Must pass a dementia screening.

Exclusion Criteria:

* Parkinson's, Alzheimer's disease, or any other neurodegenerative disease
* Terminal illness
* Severe motor impairment
* Not living in the Tallahassee area for the entire 6 month study period

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Three-Item Loneliness Scale | Assessed at baseline and at the end of the 2-months of training
  The Three-Item Loneliness Scale was developed by Hughes et al. (https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2394670/). The minimum value is 3. The maximum value is 9. Higher scores mean more loneliness.

SECONDARY OUTCOMES:
Adherence (session number) | 2 months
  Number of sessions over 2 months
Adherence (session length) | 2 months
  Number of sessions reaching at least 80% of the assigned session duration over 2 months
General Self-Efficacy (predictor of adherence) | Assessed at baseline, predicting adherence variables over 2 months
  The 10-item General Self-Efficacy Scale (GSE) was developed by Ralf Schwarzer & Matthias Jerusalem (http://userpage.fu-berlin.de/~health/engscal.htm). The minimum value is 10. The minimum value is 40. Higher scores mean higher general self-efficacy.
Perceived Training Efficacy (predictor of adherence) | Assessed at baseline
  The 7-item Cognitive Training Belief Scale (NICT scale) measures perceived usefulness of brain training. It was developed by Rabipour & Davidson in 2015 (https://pubmed.ncbi.nlm.nih.gov/25591472/). The minimum value is 7. The maximum value is 49. High scores mean higher expectations of brain training efficacy.
Self-Efficacy of Cognitive Training (predictor of adherence and training outcome) | Assessed at baseline and at the end of the 2-months of training
  The 12-item Self-Efficacy of Cognitive Training is a composite measure of self-efficacy of cognitive training based on the Health Belief Model. The minimum value is 12. The maximum value is 84. Higher scores mean lower confidence in computerized cognitive training.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe He, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No